CLINICAL TRIAL: NCT05808504
Title: Investigation of the Benefits of Electrical Non-invasive Stimulation on Cognitive Symptoms in Parkinson's Disease
Acronym: STIMPARK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: C21-76; 2022- A00767-36 (Registry Identifier: IDRCB)
Record Dates: First submitted 2023-03-13; First posted 2023-04-11 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Parkinson Disease
Keywords: Transcranial alternating current stimulation; Inhibition; Cognitive symptom; High resolution encephalography; Parkinson disease
MeSH Terms: conditions — Parkinson Disease; Inhibition, Psychological; Neurobehavioral Manifestations | interventions — Neuropsychological Tests; salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: The experimental phase will consist of 3 visits. A first one will consist of a neuropsychological exam with the MoCA, STAI, MADRS and LARS scales. Participants will also perform the Stop Task with an EEG recording. V1 has several purposes: check for inclusion criteria, define subject-specific frequency used for the stimulation, based on EEG analysis. With V1 we will also make sure that PD patients (recruited after controls), have an impaired performance at the task compared to controls. After V1, two other visits will be carried out with a 3 month interval. At V2, participants will be offered in a pseudo-randomized order either the real stimulation or the sham stimulation, with inhibition and EEG assessment (total time 45 min) before and after stimulation. The stimulation condition will be reversed during V3. V2 or V3 will also be accompanied by a brief neurological exam using the Hoehn and Yahr, and Schwab and England evaluations, and a measure of the levodopa equivalent daily dose.
Who Masked: Participant, Care Provider
Masking Description: Sham and real tACS will be applied with the same equipment (StarStim, Neuroelectrics). The stimulation will consist in applying a current (max 2 mA) at frontal sites (F8 and Cz) for 12-15 minutes during the task. A 10 s ramp (fade-in/fade-out) will be used to avoid current perception of the stimulation and optimize blinding. Sham stimulation will be done using the same protocol, but with no stimulation in between onset and offset. According to the most recent literature (Russo et al., 2013), tACS does not usually cause other sensations, allowing to distinguish it from sham. EEGs will be performed with the same chronology and monitoring. As a whole V2 and V3 will consist of this pattern : task+EEG before stimulation, then task+stimulation, then task+EEG. Blinding of the experimenter will be made possible because it is the PI who will start the stimulation program and he will not be involved in the analysis of the raw data and a random number will be given to the participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients with Parkinson disease (Experimental): Patients with idiopathic PD. Will receive real or sham transcranial alternating current stimulation at the second visit according to the randomization order. The other stimulation condition will be applied at the third visit.
  Interventions: Other: Neuropsychological assessment; Other: Neurological assessment; Other: Cognitive task; Procedure: EEG; Procedure: tACS (real or sham)
- Healthy volunteers (Experimental): Healthy volunteers with no major cognitive impairment. Will receive real or sham transcranial alternating current stimulation at the second visit according to the randomization order. The other stimulation condition will be applied at the third visit.
  Interventions: Other: Neuropsychological assessment; Other: Cognitive task; Procedure: EEG; Procedure: tACS (real or sham)

INTERVENTIONS:
Other: Neuropsychological assessment — interview with a neuropsychologist and carrying out tests measuring overall cognitive abilities, depression, apathy and anxiety (respectively using the MOCA, MADRS, LARS, STAI scales)
Other: Neurological assessment — Only for patients with Parkinson disease. Evaluation consisting in a disease severity assessment using the Hoehn and Yahr and Schwab and England scales, as a well as a measure of levodopa equivalent daily dose.
  Arms: Patients with Parkinson disease
Other: Cognitive task — The task consists in pressing a left or right button as fast and as accurately as possible according to the direction of an arrow displayed at the center of a screen. On 25 % of the trials, a "stop" signal will occur right after the stimulus, indicating the participant to stop his impending button press. The delay between the presentation of the arrow stimulus and the stop signal will be adjusted to ensure a final 50% accuracy (decreased following an accurate response and increased after an error), which is necessary to comply with the assumptions for a robust calculation of the stop signal reaction time (SSRT).
Procedure: EEG — A high-resolution (256 channels) electroencephalographic recording will be done at rest and during the Stop task, before and after each real or sham stimulation.
Procedure: tACS (real or sham) — Real or sham tACS will be applied with the same equipment (StarStim, Neuroelectrics). The stimulation will consist in applying a current (max 2 mA) at frontal sites (F8 and Cz according to standard EEG position, and defined based on dosimetry analyses on averaged head models) for 12-15 minutes during the task. A 10 s ramp (fade-in/fade-out) will be used to avoid current perception of the stimulation and optimize blinding. Sham stimulation will be done using the same protocol, but with no stimulation in between onset and offset.

SUMMARY:
Parkinson's disease is the second most common neurodegenerative disease after Alzheimer's disease.

It is mostly characterized by the presence of motor difficulties. However, it can also be accompanied by cognitive disorders which have an equally significant impact on the quality of life of patients and which are not relieved by any treatment.

Among the functions affected by Parkinson's disease, inhibition is an essential process for adapting our behaviors in daily life. Inhibition allows us to stop an action that is no longer required or appropriate to the situation in which we find ourselves in. For example, it comes into play when we have to stop at a "stop" sign while driving.

Recent studies suggest that it could be possible to improve the functioning of these processes by using non-invasive brain stimulation tools. Transcranial alternating current electrical stimulation has thus showed promising results in improving functions such as working memory. This technique is completely painless and non-invasive and consists in applying an electric current of very low intensity (barely perceptible) at the level of the scalp, using electrodes.

The investigators are conducting a study to test whether transcranial alternating current electrical stimulation could improve the functioning of the inhibition process which is altered in patients. For this, the investigators will measure this process using a task performed on a computer (the Stop Signal Reaction Time Task), as well as brain activity using a method called "electroencephalography", before and after stimulation. For this study, the investigators will include 50 patients and 40 healthy participants to investigate the effect of the stimulation on inhibition.

ELIGIBILITY:
Inclusion Criteria:

For all participants:

* Affiliation to a social security scheme or beneficiary of such a scheme.
* Age over 18 years old.
* Age less than 75 years old
* Correct or correctly corrected view (on simple declaration by the patient).
* Subject having received information on the protocol and having provided informed and written consent to participate.

Criteria exclusive to patients:

- Idiopathic Parkinson's disease according to United Kingdom Parkinson's criteria Brain Bank disease (Hughes et al., 1992).

Exclusion Criteria:

For all participants:

* Major cognitive impairment (Moca < 22) or severe neurocognitive disorder according to DSM-V (Diagnostic and statistical manual of mental disorders -V);
* Motor difficulties preventing the achievement of the task.
* Drug or alcohol addiction.
* Adult subject to legal protection (safeguard of justice, curatorship, guardianship), persons deprived of liberty.
* Present or past moderate to severe psychiatric pathology (obsessive compulsive, bipolar disorder, schizophrenia, etc.).
* Potential for pregnancy or confirmed pregnancy. A pregnancy test will be performed on inclusion.for women of childbearing age.

Criteria exclusive to patients:

* Present or past neurological pathology other than Parkinson's disease (accident stroke, head trauma, etc.).
* Deep brain stimulation treatment.

Exclusive to healthy participants:

- Present or past neurological pathology.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-05-03 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Difference in cognitive performance measured by the stop signal reaction time (SSRT) compared between real and sham stimulation conditions | 5 months

SECONDARY OUTCOMES:
The difference in the dynamic changes in functional networks during the task between real and sham stimulation. | 5 months
  The difference in the dynamic changes in functional networks during the task between real and sham stimulation measured by the averaged lifespan (in ms) if the networks identified with the weighted phase lag index.
The difference in network parameters derived from graph theory between real and sham stimulation. | 5 months
  The difference in network parameters derived from graph theory between real and sham stimulation. measured by the functions of the brain connectivity toolbox (matlab) : degree distribution, path length, betweenness centrality, clustering coefficient.
The existence of correlations between the changes in network measures between real and sham stimulation mentioned above and the behavioral differences measured between real and sham stimulation. | 5 months
  Correlations will be calculated in R using the spearman rank correlations between (i) changes in network measures between real and sham stimulation : averaged network lifespan, degree distribution, path length, betweenness centrality, clustering coefficient, and (ii) behavioral differences in SSRT (ms).

CONTACTS AND LOCATIONS:
Overall Officials: Paul Sauleau, MD, Principal Investigator — Rennes University Hospital
Locations (1):
- CHU de Rennes, Rennes, France

IPD SHARING:
Plan to Share IPD: No